CLINICAL TRIAL: NCT05981378
Title: Genomic Approaches to Dissect Human Host-pathogen Interactions in the Amazonian Rainforest
Acronym: PATHO-NAT
Status: Not yet recruiting | Type: Observational
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: Institut Pasteur (Industry)
Responsible Party: Sponsor
Other Study IDs: 210828
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Host-Pathogen Interactions
Keywords: Tropical Rainforest; Genomics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, serum, plasma, saliva, feces, peripheral blood mononuclear cells,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Native Amazonian group: Amazonian people that belongs to a indigenous community located in the Peruvian Amazon
- Urban Amazonian mestizos group: Amazonian mestizo people that lives on a urban district in the Peruvian Amazon

SUMMARY:
This observational study, aims to characterize with a multi-omic approach, the impact of host genetics and the pathogenic environment on immune response variation in Native Amazonians in comparison with Mestizo Amazonian, a severely underrepresented population in genomic studies.

Various samples will be taken from the participants, including blood, urine, saliva, etc. From the blood sample, peripheral blood mononuclear cells will be obtained and will give us information about the differences between immune response variation of Amazonian population. From the other samples we will be able to obtain additional information on the risk factors related to the difference in the immune response of the participants.

DETAILED DESCRIPTION:
The Amazon rainforest is characterized by adverse climatic conditions and a great diversity of pathogenic microorganisms that, consequently, would generate a selective pressure on the human immune response with a high impact on mortality. Some of the best characterized examples of human genetic adaptation have been related to infections; for example, the alleles causing sickle cell anemia, thalassemia and malaria. In addition, the introduction of infectious diseases from the "old world" during Spanish colonization in the 15th century and the urbanization of the last few centuries in the Amazon has also generated rapid adaptation that could drive variation in immune response. However, the evolutionary mechanisms that contributed to the adaptation of human defense against the aforementioned phenomena and events in this region are poorly understood. For this reason, studying these human genetic mechanisms in native populations would allow us to identify new genes that would be associated with resistance to infections, and also to explore the signs of rapid adaptation to the environment to which Amazonian populations have been exposed throughout their history.

We propose to study the variation of the immune system in Amazonian populations, studying together the degree of diversity with different approaches: genomic, epi-genomic and transcriptomic of the host and viral exposome, taking into consideration sociodemographic characteristics and comorbidities, which may shape the immune response. This study will provide new insights into variants in the human genome that affect the immune response, thereby increasing our understanding of the etiology and susceptibility to immune-related diseases, mainly tropical infectious diseases. Because human genetic studies are underrepresented in Native American populations, the knowledge gained would reduce the existing inequality in health knowledge between Native and non-Native populations.

ELIGIBILITY:
Inclusion Criteria:

* People over 18 years of age who agree to participate in the study and sign the informed consent
* People whose parents and grandparents were born in the Peruvian Amazon.
* For volunteers from native communities, whose parents and grandparents belong to the same native community.

Exclusion Criteria:

* People who do not wish to have 40 mL of blood taken
* People who are passing through a febrile illness (fever during the last 5 days to the date of enrollment).
* Pregnant women
* People over 65 years old
* Breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Amazonian Peruvian Native American and Amazonian mestizo population between 2023-2024
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-08-02 (Estimated); Primary Completion 2024-11-20 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Genes showing different transcriptional profiles and methylation pattern according environment, genetic ancestry and past viral exposure | Baseline
  We will measure genome-wide expression profiles in peripheral blood mononuclear cells after stimulation for 6 hours with: (i) dengue virus, a major public health burden in the region, (ii) gardiquimod, an imidazoquinoxaline compound that activates toll like receptor 7/toll like receptor 8, able to sense viruses and intracellular pathogens; and (iii) lipopolysaccharide, a toll like receptor 4 agonist, to obtain a general view of responses to viruses and bacteria.
  Gene expression profiles will be measured using RNA-seq.
Genetic and epigenetic diversity of amazonian population | Baseline
  Using saliva from participants as source of DNA, we will perform whole-genome sequencing (WGS) at 8-10xcoverage.
Impact of microbial exposures on immune response | Baseline
  The viral exposome will be characterized in the 300 donors using a new tool call "VirScan", which identifies antibodies against >600 pathogens and allergens, including viruses (>1,200 viral strains) that are highly prevalent in the Amazonian, such as dengue, hepatitis B/C/D, or Mayaro virus.
Genetic variants associated wit transcriptional response to immune activation and DNA methylation variation | Baseline
  We will assess the host genetic factors controlling transcriptional responses and methylated DNA levels by mapping expression and methylation quantitative trait loci (eQTL and methylated eQTLs, respectively).

SECONDARY OUTCOMES:
Demographic and admixture history of amazonian population | Baseline
  Using saliva from participants as source of DNA, we will perform whole-genome sequencing (WGS) at 8-10xcoverage.
Natural selection role in shaping immune response variation in Amazonians | Baseline
  We will employ an enrichment approach to test whether eQTLs, associated to specific cell-types or conditions, have been preferentially targeted by selection.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Web page of the ethical review board of Universidad Peruana Cayetano Heredia — https://investigacion.cayetano.edu.pe/duari/ciei/
- Available data/document: Study Protocol — https://drive.google.com/drive/folders/1SJk21vz3MOlaF8tSVnwPlwo9sxmmewZp?usp=drive_link — Google drive link to visualize the study protocol in Spanish and English